CLINICAL TRIAL: NCT05656729
Title: Studio Clinico Randomizzato in Doppio Cieco, Controllato Verso Placebo, a Gruppi Paralleli, Sull'efficacia Clinica Di Un Prodotto a Base Di Probiotici Nel Migliorare I Comuni Sintomi Da Raffreddamento E La Risposta Immunitaria in Adulti Sani - ImmunoCold 2021
Brief Title: Effect of a Multistrain Probiotic on Cold Symptoms in Healthy Patients with an History of Upper Airways Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Giacomo Caio, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ImmunoCold 2021
Record Dates: First submitted 2022-12-05; First posted 2022-12-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-04

CONDITIONS: Cold Symptom
Keywords: cold; cold symptoms; probiotics
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 8-week daily administration
  Interventions: Dietary Supplement: Placebo
- Multistrain probiotic (Active Comparator): Dietary Supplement: Multistrain Probiotic 12-week daily administration
  Interventions: Dietary Supplement: DefensePlus

INTERVENTIONS:
Dietary Supplement: DefensePlus — Multistrain probiotic:L. plantarum PBS077, L. acidophilus PBS066, B. lactis BL050, Maltodextrins, Vitamin B12, Vitamin, B6 Folic acid, Magnesium, silicon dioxide
  Arms: Multistrain probiotic
Dietary Supplement: Placebo — Maltodextrins, Vitamin B12, Vitamin, B6 Folic acid, Magnesium, silicon dioxide
  Arms: Placebo

SUMMARY:
The study is a double-blind randomized clinical trial which aims to evaluate the efficacy of a multi strain probiotic in human adults in controlling and improving cold symptoms and inflammatory response

DETAILED DESCRIPTION:
Adult subjects (age 18-44) with a history of upper airways infection, will be assigned to placebo or probiotic groups and take either placebo or probiotic dietary intervention for 12 weeks. After that, a 6 weeks follow-up. The answers at: Common Cold Questionnarie (CCQ), Wisconsin Upper Respiratory Symptoms Survey-21 (WURSS-21) and quality of life score (SF-36) will be compared in the two groups. In addition, serological markers (blood count, lymphocyte subpopulation (B, T, T4, T8, NK), IFN-γ and IL-10 levels) will be evaluated over a 18 week period.

ELIGIBILITY:
Inclusion Criteria:

people who:

* are willing and capable of joining the study
* are willing of not varying their routine (lifestyle, physical activity..) during the study
* are willing of not varying their diet during the study
* are willing of using only the testing product during the study
* are willing of not using products that may interfere with the testing product
* have not recently joined similar studies
* have signed informed consent

Exclusion Criteria:

subjects:

* not filling the inclusion criteria
* with suspected or confirmed sensibility to one or more product component
* with chronic diseases (cardiovascular congenital diseases, hepatic diseases, renal disease, immunodeficiency)
* undergoing antibiotic/pharmacological treatment
* with other concomitant disease (infective, respiratory, gastrointestinal, immune)
* who underwent an immunomodulating treatment in the past 4 weeks
* who underwent an immunosuppressant therapy in the past 3 months
* with severe disease ongoing
* who abuse of alcohol and/or drugs
* who are considered not eligible by the investigator
* not able to communicate due to language barriers, mental issues or cerebral functioning impairment

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Cold symptoms evaluation | 18 weeks
  Cold symptoms will be evaluated before and after treatment through Common Cold Questionnaire(CCQ). Highest score: 27, Lowest 0. Higher scores indicate worst symptoms

SECONDARY OUTCOMES:
Change of Wisconsin Upper Respiratory Symptoms Survey (WURSS-21) | 18 weeks
  Changes of WURSS-21 questionnaire will be assessed before and after treatment. Highest score: 147, Lowest 0. Higher scores indicate worst symptoms
Change of Short Form Health Survey 36 (SF-36) | 18 weeks
  Higher score on Short Form Health Survey 36 (SF-36) questionnaire will be considered as an improvement of life quality. Highest score: 147, Lowest 0. Higher scores indicate better perception of one's health
Inflammatory status | 18 weeks
  A reduction of inflammatory markers (INF-y, IL-10, and lymphocite B, T, T4, T8, NK) will be considered as an improvement of inflammatory status

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria di Ferrara, Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No